CLINICAL TRIAL: NCT01746160
Title: A Short-term Longitudinal Follow-up After C1 Implant Stability Values.
Brief Title: Longitudinal Follow-up After C1 Implant Stabilization Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C1implantstability-HMO-CTIL
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2016-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: dental implant; healing; implant stability
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- C1 Implant (Experimental): Patient having C1 implant installed.
  Interventions: Drug: C1 Implant

INTERVENTIONS:
Drug: C1 Implant — Patients treated with dental implants.
  Other Names: Treated patients; Implant cases

SUMMARY:
The aim of the study is to describe the changes found in C1 dental implants through their early healing period.

Patients requiring a standard installation of one or two implants in the maxilla, without any need for bone augmentation, will be frequently followed for 90 days. In every meeting the implants' ISQ values (values denoting the implant stability as being measured by a dedicated, commercially available, appliance called 'Osstell').

The implants' measured ISQ values will be used to describe the changes that may be found in the implants' stability through their healing period.

At the end of the study the patients will be referred to their treating doctor for the completion of implants' restoration (i.e. crown).

DETAILED DESCRIPTION:
10 Patients requiring standard implant installation in their maxilla will be recruited to the study.

Inclusion criteria:

* Men and women over the age of 18.
* The patient will be willing, and will be available to attend all the follow-up meetings.
* The patient will accept and sign an informed consent form before the beginning of the study.

Exclusion criteria:

* Pregnant women or women who are breast feeding.
* Patient suffering of untreated periodontal disease.
* Patient who smoke more than 10 cigarettes per day.
* Alcohol abuse.
* Patient suffering of either uncontrolled Diabetes, Osteoporosis, rheumatic arthritis, neoplastic or pre-cancerous condition, or any other condition limiting standard implant installation procedure.
* Patient who need some bone augmentation prior.
* Immediate implant placement or restorations.

Course of study:

Every patient found eligible to the study will need to go through a CT scan of the implantation site (as required).

Before the operation 2 gr of AMOXICILLIN (or 600mg of CLYNDAMYCIN - in case of allergy) will be administered. The implants will be installed in a standard approach under local anesthesia, as customary being done. The implants' installation torque will be recorded.

At the end of the operation the patients will be instructed to rinse their mouth with Chlorhexidine solution for one week.

Eventually the implants will be restored and loaded after the common 3 months healing period.

Follow-up appointments:

The patients will be monitored through a period of 3 months. The patients will be instructed to return to a follow-up examination 2, 4, 7, 14, 21, 28, 45, 60 and 90 days after the operation. On each meeting the implants' ISQ values will be measured using an 'Osstell' appliance.

An x-ray intra-oral radiogram will be taken right after the end of the operation and at the end of the follow-up (i.e day 90).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18.
* The patient will be willing, and will be available to attend all the follow-up meetings.
* The patient will accept and sign an informed consent form before the beginning of the study.

Exclusion criteria:

* Pregnant women or women who are breast feeding.
* Patient suffering of untreated periodontal disease.
* Patient who smoke more than 10 cigarettes per day.
* Alcohol abuse.
* Patient suffering of either uncontrolled Diabetes, Osteoporosis, rheumatic arthritis, neoplastic or pre-cancerous condition, or any other condition limiting standard implant installation procedure.
* Patient who need some bone augmentation prior.
* Immediate implant placement or restorations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in implant ISQ value. | 90 days (at end of the follow-up).
  The change in implants' stability values that were measured by an 'Osstell' appliance at the end of the study as compared to their baseline value.

SECONDARY OUTCOMES:
Implant Marginal Bone Loss (MBL). | 90 days (At the end of the follow-up).
  The amount of the marginal bone loss (MBL) as measured by comparing two intra-oral radiogram taken right after the operation and at the end of the follow-up period.

OTHER OUTCOMES:
Implant survival rate. | 90 days (At the end of the follow-up).
  The rate of the implants found to be integrated at the end of the study (100% is anticipated).

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Lemberg, PhD, Principal Investigator — IRB coorinator
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Nedir R, Bischof M, Szmukler-Moncler S, Bernard JP, Samson J. Predicting osseointegration by means of implant primary stability. Clin Oral Implants Res. 2004 Oct;15(5):520-8. doi: 10.1111/j.1600-0501.2004.01059.x. PMID 15355393
- [Background] Glauser R, Sennerby L, Meredith N, Ree A, Lundgren A, Gottlow J, Hammerle CH. Resonance frequency analysis of implants subjected to immediate or early functional occlusal loading. Successful vs. failing implants. Clin Oral Implants Res. 2004 Aug;15(4):428-34. doi: 10.1111/j.1600-0501.2004.01036.x. PMID 15248877
- [Background] Turkyilmaz I, Sennerby L, Tumer C, Yenigul M, Avci M. Stability and marginal bone level measurements of unsplinted implants used for mandibular overdentures: a 1-year randomized prospective clinical study comparing early and conventional loading protocols. Clin Oral Implants Res. 2006 Oct;17(5):501-5. doi: 10.1111/j.1600-0501.2006.01261.x. PMID 16958688
- [Background] Hobkirk JA, Wiskott HW; Working Group 1. Biomechanical aspects of oral implants. Consensus report of Working Group 1. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:52-4. doi: 10.1111/j.1600-0501.2006.01358.x. PMID 16968381
- [Background] Aparicio C, Lang NP, Rangert B. Validity and clinical significance of biomechanical testing of implant/bone interface. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:2-7. doi: 10.1111/j.1600-0501.2006.01365.x. PMID 16968377